CLINICAL TRIAL: NCT01784731
Title: Brugerbetaling i Almen Praksis (In Danish: User Charges for General Practitioner Services)
Brief Title: User Charges for General Practitioner Services in Denmark
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Christian Kronborg, Associate professor, University of Southern Denmark
Other Study IDs: SDU1
Record Dates: First submitted 2013-02-04; First posted 2013-02-06 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Consequences of User Charges

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients
  Interventions: Behavioral: Willingness to pay

INTERVENTIONS:
Behavioral: Willingness to pay

SUMMARY:
Currently, office visits at general practitioners is free of charge for patients. However, public commissions and the Danish Economic Council have suggested to implement user charges for services that currently is free of charge. The aim of this study is to examine the consequences of introducing user charges for general practitioner services. Data for the project will be collected from patients who have an appointment with a general practitioner. Patients will be asked whether they are willing to pay a specified amount for the consultation that they have scheduled. After the consultation, the GP register diagnoses.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an appointment for a visit in a general practitioner clinic
* Reads and understand Danish

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients enrolled with a general practitioner clinic
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2013-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Willingness to pay | once
  Whether a patient accept a specified amount for a GP consultation

SECONDARY OUTCOMES:
Diagnoses | Once
  Diagnoses according to the Danish version of the International Classification of Primary Care (ICPC9

CONTACTS AND LOCATIONS:
Locations (1):
- Lægerne Nyenstad, Nyborg, Denmark

REFERENCES:
- [Derived] Kronborg C, Pedersen LB, Fournaise A, Kronborg CN. User Fees in General Practice: Willingness to Pay and Potential Substitution Patterns-Results from a Danish GP Patient Survey. Appl Health Econ Health Policy. 2017 Oct;15(5):615-624. doi: 10.1007/s40258-017-0325-y. PMID 28364368